CLINICAL TRIAL: NCT00331318
Title: Encoding a Motor Memory Through Metaplasticity
Brief Title: Improving Hand Movement Training Through Electrical Stimulation of the Brain
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060171; 06-N-0171
Record Dates: First submitted 2006-05-27; First posted 2006-05-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Metaplasticity
Keywords: Transcranial Direct Current Stimulation (tDCS); Transcranial Magnetic Stimulation (TMS); Motor Learning; Brain Plasticity; Healthy Volunteer; HV

SUMMARY:
This study will determine if applying electrical stimulation of the brain can influence training to perform finger movements. The study may provide information that can be used to design rehabilitation therapies for people who have lost the ability to move a part of their body, such as an arm, leg, or hand following a stroke.

Healthy volunteers 18-50 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, MRI (if one has not been done within the last year), questionnaire to evaluate memory and attention and a pregnancy test for women who can become pregnant.

Participants have the following tests and procedures in seven sessions over about 8 weeks:

* Questionnaires to test attention, fatigue and mood before, during and after each session
* Surface electromyography: Electrodes are filed with a conductive gel and taped to the skin over one small hand muscle to measure the electrical activity of muscles.
* Transcranial magnetic stimulation: A wire coil is held on the scalp. A brief electrical current passes through the coil to stimulate the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil.
* Transcranial direct stimulation (tDCS) before and during motor training: Small, wet sponge electrodes are applied to the head - one above the eye and the other on the back of the head. A small electrical current is passed between them. The subject may feel an itching or tingling sensation under the electrodes or see light flashes.
* Motor learning under tDCS: tDCS is repeated while the subject performs the training task. The training task consists of performing voluntary brisk thumb movements in a direction opposite to TMS-induced movement directions, during 30 minutes. Training blocks are in 10-minute segments and tDCS is applied during the first 20 minutes.
* Behavioral measurements: Evaluation of learned movement tasks.

DETAILED DESCRIPTION:
OBJECTIVES:

Training leads to performance improvements and motor learning. Cortical plasticity associated with training (use-dependent plasticity, UDP) contributes to performance improvements after brain lesions such as stroke. Recently, several interventional strategies have been proposed to enhance UDP, including pharmacological approaches and brain stimulation. The magnitude of improvements identified with these techniques is limited. It would be very useful to enhance UDP beyond the limited effects of previously proposed interventions.

One strategy recently proposed to enhance the effect of brain stimulation techniques on the cerebral cortex is metaplasticity. This strategy focuses on the purposeful manipulation of cortical activity before applying brain stimulation. For example, previous work demonstrated that the magnitude of increase in cortical excitability elicited by stimulation of the primary motor cortex (M1) is more prominent if stimulation is applied on a hypoactive M1. An initial down-regulation of M1 activity (i) amplifies the effect of a subsequent intervention that increases M1 activity, and (ii) reduces inter-individual variability.

It is unknown if this metaplasticity strategy can enhance the beneficial effects of anodal tDCS (tDCS anodal) on training effects as it does with cortical excitability, an issue of scientific and clinical interest, and the overall hypothesis of this protocol.

Here, we will test the hypothesis that metaplasticity (tDCS cathodal) followed by tDCS anodal plus motor training will result in more prominent UDP than control interventions.

STUDY POPULATION

6 healthy adult volunteers for parameters estimation plus 25 healthy adult volunteers (total = 31 healthy adult volunteers)

DESIGN

In this protocol, down-regulation of M1 activity will be accomplished by applying tDCS cathodal, a tool extensively described in the literature to induce this effect. Therefore, we will test the effects of this metaplasticity intervention on the beneficial action of tDCS anodal to M1 in combination with motor training (MT). After a familiarization session, subjects will participate in 6 randomized sessions in a cross-over design:

1. Preconditioning tDCS cathodal followed by Intervention tDCS anodal plus MT Purpose Target metaplasticity condition
2. Preconditioning Sham followed by Intervention Sham plus MT Purpose Effects of motor training alone
3. Preconditioning Sham followed by Intervention tDCS anodal plus MT Purpose Mild improvement in training effects
4. Preconditioning tDCS cathodal followed by Intervention Sham plus MT Purpose Effects of tDCS cathodal alone on MT
5. Preconditioning tDCS anodal followed by Intervention Sham plus MT Purpose Effects of polarity on tDCS effects
6. Preconditioning tDCS anodal followed by Intervention tDCS anodal plus MT Purpose Control for the metaplasticity condition

MT will consist of brisk repetitive thumb movements in a direction opposite to the baseline direction of thumb movements evoked by focal transcranial magnetic stimulation (TMS), in a well-characterized UDP protocol.

The primary outcome measure reflecting the encoding of a motor memory will be the increased proportion of TMS-evoked movements falling within the target training zone (TTZ) as a function of MT and metaplasticity interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* age between 18-50 years
* able to perform tasks required by the study
* willing and able to give consent
* willing to make an eight-week commitment to the study
* possibility of obtaining TMS-evoked thumb movements in a consistent direction at baseline

EXCLUSION CRITERIA:

* unable to perform the tasks
* history of severe alcohol or drug abuse, psychiatric illness such as severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score (MMSE) of 23 or less), or degenerative brain processes such as Alzheimer's disease
* severe uncontrolled medical problems (e.g., cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others), more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease
* problems with movement of the hands
* receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants (for the TMS component)
* pregnancy and during lactation
* medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., dental braces, pacemakers, implanted medication pumps, cochlear devices, neural stimulators, metal in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31
Dates: Start 2006-05-24; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Siebner HR, Lang N, Rizzo V, Nitsche MA, Paulus W, Lemon RN, Rothwell JC. Preconditioning of low-frequency repetitive transcranial magnetic stimulation with transcranial direct current stimulation: evidence for homeostatic plasticity in the human motor cortex. J Neurosci. 2004 Mar 31;24(13):3379-85. doi: 10.1523/JNEUROSCI.5316-03.2004. PMID 15056717